CLINICAL TRIAL: NCT03899532
Title: The Effect of Remote Ischemic Conditioning (RIC) on Inflammatory Biomarkers and Outcomes in Patients With TBI
Brief Title: Remote Ischemic Conditioning in Traumatic Brain Injury
Acronym: MOTION
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No eligible participants were enrolled.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1901298756
Record Dates: First submitted 2019-03-27; First posted 2019-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2022-05

CONDITIONS: Traumatic Brain Injury; Brain Injuries; Brain Trauma; Brain Injuries, Traumatic
Keywords: Remote Ischemic Conditioning; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Remote Ischemic Conditioning (Experimental): Remote ischemic conditioning will be performed using a standard manual blood pressure cuff. The pressure in the blood pressure cuff will be maintained at 30 mm of Hg higher than the patient's systolic blood pressure. 4 cycles of ischemic conditioning will be performed each day for a period of 7 days. Each cycle consists of 5 min of controlled upper limb ischemia (cuff up) followed by 5 min of reperfusion (cuff down). The total duration of the treatment cycle will be 40 min. The study protocol is based on our published literature in traumatic brain injury.
  Blood samples will be collected at 0 hours (before randomization). Then the first 4 cycles of RIC (done consecutively) will be performed, blood samples will be taken at 6 hours post randomization and then at 24 hours post randomization. RIC cycles will then be performed on a daily basis followed by taking a blood sample once daily during the patients' length of stay up to a maximum of 7 days
  Interventions: Device: Remote Ischemic Conditioning
- No Remote Ischemic Conditioning (Placebo Comparator): Blood samples will be collected at 0 hours (before randomization). Blood samples will then be collected at 6 hours post randomization and 24 hours post randomization. These patients will not receive daily RIC therapy but will only have their blood drawn once daily during the patients' length of stay up to a maximum of 7 days.
  Interventions: Other: No-Remote Ischemic Conditioning

INTERVENTIONS:
Device: Remote Ischemic Conditioning — Standard manual blood pressure cuff
  Arms: Remote Ischemic Conditioning
Other: No-Remote Ischemic Conditioning — No-Remote Ischemic Conditioning
  Arms: No Remote Ischemic Conditioning

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of death among trauma patients accounting for one-third of all trauma mortalities. Patients who survive the initial trauma are liable to secondary insults from the ensuing inflammatory state in the brain. Treatment goals are aimed at reducing secondary injury. Maintaining adequate brain perfusion, limiting cerebral edema, and optimizing oxygen delivery are part of established treatment protocols. Numerous therapeutics have been evaluated as potential treatment for TBI with very limited success and there is no medication that alters survival.

Various novel therapeutic options have been investigated to prevent the secondary brain injury. Remote Ischemic Conditioning (RIC) is one of these therapies. RIC involves decreasing blood flow to a normal tissue usually the arm by inflating the blood pressure cuff 30mmHg over the systolic blood pressure. The decreased blood flow or ischemia is maintained for 5 minutes followed by releasing the pressure and re-perfusion of the arm. This cycle is usually repeated 4 times. RIC has been shown to improve outcomes in patients with heart attacks, strokes, elective neurosurgeries.

A prospective observational study and a randomized clinical trial has shown the protective effect of RIC in TBI patients. Additionally, multiple studies in animals have shown that RIC is neuroprotective after TBI. RIC is non-invasive and harmless except for a little discomfort in the arm. The aim of the study is to evaluate the impact of RIC on long term outcomes in patients with TBI.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) remains one of the leading causes of death and disability in the United States. Secondary brain injury caused by the complex interplay of inflammatory mediators induced by a primary insult is the major contributing factor for morbidity and mortality after TBI. While the primary injury is irreversible, the inflammatory cascade leading to the development of the secondary injury may be preventable. As a result, all the current research in TBI is focused on preventing initiation of this secondary insult.

Remote ischemic conditioning (RIC) is a process where normal tissues are subjected to short cycles of ischemia and reperfusion, which have been shown to reduce the sequelae of an ischemic injury at a remotely injured site. RIC has been shown to improve the outcomes after myocardial infarction, sepsis, transplantation, reimplantation, and elective neurologic surgery.It is thought to work by releasing endogenous systemic anti-inflammatory mediators and humoral factors and by using neural pathways, rendering global protection to the body against subsequent ischemic insults in a remote are. This protection provided by RIC has two phases, an early (short) phase and a late (prolonged) phase, both of which have proven to be effective in reducing ischemic size and improving survival. Multiple animal studies and a small randomized clinical trial have shown the protective effect of RIC in patients with TBI. The effectiveness of RIC in patients with traumatic brain injury is still under investigation not yet established.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 17years.
2. Diagnosis of traumatic brain injury.
3. Glasgow Coma Scale (GCS) ≤13
4. Intra-cranial hemorrhage (ICH) on initial brain CT scan

Exclusion Criteria:

1. Patients with traumatic brain injury >24 hours
2. Transferred from other centers
3. Declined to participate in the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in the level of Inflammatory Biomarkers (pg/ml) | Before randomization, 6 hours post randomization, 24 hours post randomization, once daily during the patients' length of stay up to a maximum of 7 days afterwards
  Level of tumor necrosis factor alpha (TNF-alpha), Level of interleukin 1 (IL-1),Level of interleukin 6 (IL-6), Level of interleukin 8 (IL-8), and Level of interleukin 10 (IL-10).
Change in the level of C-reactive protein C-reactive Protein mg/dl | Before randomization, 6 hours post randomization, 24 hours post randomization, once daily during the patients' length of stay up to a maximum of 7 days afterwards
  C-reactive protein
Change in the Level of pro-calcitonin (ng/ml) | Before randomization, 6 hours post randomization, 24 hours post randomization, once daily during the patients' length of stay up to a maximum of 7 days afterwards
  Level of pro-calcitonin
Change in the Level of cardiac biomarker: Troponin c (ng/ml) | Before randomization, 6 hours post randomization, 24 hours post randomization, once daily during the patients' length of stay up to a maximum of 7 days afterwards
  Troponin c
Change in the Level of cardiac biomarker: Creatinine Phosphokinase (ug/ml) | Before randomization, 6 hours post randomization, 24 hours post randomization, once daily during the patients' length of stay up to a maximum of 7 days afterwards
  Creatinine Phosphokinase
Change in the Level of cardiac biomarker: Creatine Kinase MB CKMB (ug/ml) | Before randomization, 6 hours post randomization, 24 hours post randomization, once daily during the patients' length of stay up to a maximum of 7 days afterwards
  Creatine Kinase MB

SECONDARY OUTCOMES:
Discharge Disposition/Destination | Last hospitalization day
Mortality | Last hospitalization day, 30 days post-discharge
Glasgow Outcome Scale-Extended (points) | Last hospitalization day, 30 days
  Functional independence level assessment: The Extended Glasgow Outcome Scale (GOSE) is a global scale for functional outcome that rates patients into eight categories. The categories of severe disability, moderate disability and good recovery are subdivided into a lower and upper category. The scale will be used to evaluate the patient's functional status
Glasgow Coma Scale (points) | Last hospitalization day, 30 days
  Neurological status assessment The Glasgow Coma Scale is divided into three components which are scored separately: ocular response (assessment 1-4 points), motor response (assessment 1-6 points) verbal response (evaluation of 1-5 points).
  Scores for each component are added together to get the total that will range between a minimum of 3 points (which corresponds to a patient who does not open his eyes and no motor response to stimulation or verbal response) and a maximum value of 15 points (corresponding to a patient with open eyes, obeying orders and maintaining a consistent language).
  It has been considered that the GCS score between 15 and 13 points corresponds to a slight alteration of consciousness, a score of 12-9 points with moderate impairment and 8 points or less with a serious deterioration in level of consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Bellal Joseph, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CDCVTBI in the US ReportVTraumatic Brain Injury. Injury Center 2014. Available at: http://www.cdc.gov/traumaticbraininjury/tbi_ed.html#3. Accessed July 22, 2014
- [Background] Werner C, Engelhard K. Pathophysiology of traumatic brain injury. Br J Anaesth. 2007 Jul;99(1):4-9. doi: 10.1093/bja/aem131. PMID 17573392
- [Background] Stein DM, Kufera JA, Lindell A, Murdock KR, Menaker J, Bochicchio GV, Aarabi B, Scalea TM. Association of CSF biomarkers and secondary insults following severe traumatic brain injury. Neurocrit Care. 2011 Apr;14(2):200-7. doi: 10.1007/s12028-010-9496-1. PMID 21210304
- [Background] Saxena P, Newman MA, Shehatha JS, Redington AN, Konstantinov IE. Remote ischemic conditioning: evolution of the concept, mechanisms, and clinical application. J Card Surg. 2010 Jan-Feb;25(1):127-34. doi: 10.1111/j.1540-8191.2009.00820.x. Epub 2009 Jun 22. PMID 19549044
- [Background] Munk K, Andersen NH, Schmidt MR, Nielsen SS, Terkelsen CJ, Sloth E, Botker HE, Nielsen TT, Poulsen SH. Remote Ischemic Conditioning in Patients With Myocardial Infarction Treated With Primary Angioplasty: Impact on Left Ventricular Function Assessed by Comprehensive Echocardiography and Gated Single-Photon Emission CT. Circ Cardiovasc Imaging. 2010 Nov;3(6):656-62. doi: 10.1161/CIRCIMAGING.110.957340. Epub 2010 Sep 8. PMID 20826592
- [Background] Lim SY, Hausenloy DJ. Remote ischemic conditioning: from bench to bedside. Front Physiol. 2012 Feb 20;3:27. doi: 10.3389/fphys.2012.00027. eCollection 2012. PMID 22363297
- [Background] Konstantinov IE, Arab S, Kharbanda RK, Li J, Cheung MM, Cherepanov V, Downey GP, Liu PP, Cukerman E, Coles JG, Redington AN. The remote ischemic preconditioning stimulus modifies inflammatory gene expression in humans. Physiol Genomics. 2004 Sep 16;19(1):143-50. doi: 10.1152/physiolgenomics.00046.2004. Epub 2004 Aug 10. PMID 15304621
- [Background] Steiger HJ, Hanggi D. Ischaemic preconditioning of the brain, mechanisms and applications. Acta Neurochir (Wien). 2007 Jan;149(1):1-10. doi: 10.1007/s00701-006-1057-1. Epub 2006 Dec 14. PMID 17151832
- [Background] Konstantinov IE, Li J, Cheung MM, Shimizu M, Stokoe J, Kharbanda RK, Redington AN. Remote ischemic preconditioning of the recipient reduces myocardial ischemia-reperfusion injury of the denervated donor heart via a Katp channel-dependent mechanism. Transplantation. 2005 Jun 27;79(12):1691-5. doi: 10.1097/01.tp.0000159137.76400.5d. PMID 15973170
- [Background] Hu S, Dong HL, Li YZ, Luo ZJ, Sun L, Yang QZ, Yang LF, Xiong L. Effects of remote ischemic preconditioning on biochemical markers and neurologic outcomes in patients undergoing elective cervical decompression surgery: a prospective randomized controlled trial. J Neurosurg Anesthesiol. 2010 Jan;22(1):46-52. doi: 10.1097/ANA.0b013e3181c572bd. PMID 19996767
- [Background] Sahebally SM, Healy D, Coffey JC, Walsh SR. Should patients taking aspirin for secondary prevention continue or discontinue the medication prior to elective, abdominal surgery? Best evidence topic (BET). Int J Surg. 2014;12(5):16-21. doi: 10.1016/j.ijsu.2013.11.004. Epub 2013 Nov 15. PMID 24246172
- [Background] Loukogeorgakis SP, Williams R, Panagiotidou AT, Kolvekar SK, Donald A, Cole TJ, Yellon DM, Deanfield JE, MacAllister RJ. Transient limb ischemia induces remote preconditioning and remote postconditioning in humans by a K(ATP)-channel dependent mechanism. Circulation. 2007 Sep 18;116(12):1386-95. doi: 10.1161/CIRCULATIONAHA.106.653782. Epub 2007 Aug 27. PMID 17724264
- [Background] Wei M, Xin P, Li S, Tao J, Li Y, Li J, Liu M, Li J, Zhu W, Redington AN. Repeated remote ischemic postconditioning protects against adverse left ventricular remodeling and improves survival in a rat model of myocardial infarction. Circ Res. 2011 May 13;108(10):1220-5. doi: 10.1161/CIRCRESAHA.110.236190. Epub 2011 Apr 7. PMID 21474817
- [Background] Andreka G, Vertesaljai M, Szantho G, Font G, Piroth Z, Fontos G, Juhasz ED, Szekely L, Szelid Z, Turner MS, Ashrafian H, Frenneaux MP, Andreka P. Remote ischaemic postconditioning protects the heart during acute myocardial infarction in pigs. Heart. 2007 Jun;93(6):749-52. doi: 10.1136/hrt.2006.114504. Epub 2007 Apr 20. PMID 17449499
- [Background] Loukogeorgakis SP, Panagiotidou AT, Broadhead MW, Donald A, Deanfield JE, MacAllister RJ. Remote ischemic preconditioning provides early and late protection against endothelial ischemia-reperfusion injury in humans: role of the autonomic nervous system. J Am Coll Cardiol. 2005 Aug 2;46(3):450-6. doi: 10.1016/j.jacc.2005.04.044. PMID 16053957